CLINICAL TRIAL: NCT05022342
Title: A Descriptive Study of PIK3CA Mutations and Outcomes With Alpelisib in Patients With HR-positive and HER2-negative Advanced Breast Cancer (ABC)/ Metastatic Breast Cancer (MBC) in India
Brief Title: Study of PIK3CA Mutations and Effectiveness and Tolerability Outcomes of Alpelisib in Real-world
Acronym: SPEAR
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CBYL719CIN02
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: advanced breast cancer; metastatic breast cancer; PIK3CA mutations
MeSH Terms: conditions — Breast Neoplasms | interventions — Alpelisib; Fulvestrant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HR-positive HER2-negative ABC/MBC: Hormone receptor (HR)-positive and human epidermal growth factor receptor 2 (HER2)-negative advanced breast cancer (ABC)/ metastatic breast cancer (MBC) patients
- PIK3CA mutation positive: Patients with Phosphatidylinositol-4,5-Bisphosphate 3-Kinase Catalytic Subunit Alpha (PIK3CA) gene mutation positive
  Interventions: Other: alpelisib plus fulvestrant

INTERVENTIONS:
Other: alpelisib plus fulvestrant — Prospective observational study. There is no treatment allocation. Patients administered alpelisib plus fulvestrant, that have started before inclusion of the patient into the study will be enrolled.
  Groups: PIK3CA mutation positive

SUMMARY:
SPEAR is a non-interventional / observational, prospective, multicenter study planned to be conducted across ~ 30 sites in India, among HR-positive and HER2-negative ABC/MBC patients. This being a non-interventional study, no investigational drug or intervention will be administered as a part of the study participation. All the therapeutic decisions, as well as the type and timing of disease monitoring, laboratory tests or medical procedures will be at the discretion of the treating physician and upon patient's consent. No visits will be scheduled as a part of this non-interventional study, however, data by visits for variables will be collected for all the enrolled patients.

DETAILED DESCRIPTION:
Overall, this study will have 2 parts (Part A and Part B). However, it is to be noted that, these parts (Part A and Part B) are independent of each other and can run in parallel. The purpose of the Part A of study is to determine the proportion of PIK3CA mutation positive patients among the HR-positive and HER2-negative ABC/MBC diagnosed patients in India. The Part B of the study aims to evaluate the clinical effectiveness and tolerability of alpelisib plus fulvestrant among men, pre-menopausal women (ovarian ablation) or post-menopausal women who are PIK3CA mutation positive patients with HR-positive and HER2-negative ABC/MBC diagnosis among Indian population, in the real-world setting.

Part A- This will involve enrolling of approximately 1200 patients (males, post-menopausal women or pre-menopausal women who are receiving ovarian ablation) with a documented diagnosis of HR-positive HER2-negative ABC/MBC. The data on PIK3CA mutation status will be collected only for those patients who signs ICF for participation in the study. Once, patient signs ICF, their samples will be sent for PIK3CA mutation status testing, that will be performed at central laboratory and the results on mutation status will be reported to the investigator.

Part B- This part aims to enroll approximately 200 patients who are PIK3CA mutation positive. The patients enrolled into the Part B of the study can either be continued from Part A of the study or be a direct enrollment into the Part B of the study. For the patient's entering directly into Part B of the study, positive PIK3CA status should be available prior to study entry. All the patients entering into part B of the study must be alpelisib treatment naïve. The patients enrolled into Part B of the study, should have already been planned to receive treatment with alpelisib plus fulvestrant, based on their treating physician's discretion and upon patient's consent. The treatment decision by the physician are to be made independent of the patient's inclusion in this observational study. During the Part B of the study, data by visits for variables will be collected for the enrolled patients at every 3 months interval (±1 month), if feasible or until a maximum of 24 months observational period or lost to follow-up (End-of-study [EoS] assessment will be performed), or death, or disease progression, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

PART A:

1. Males (≥18 years of age), post-menopausal* females or pre-menopausal** females with ovarian ablation (as per physician decision).
2. Patients with confirmed diagnosis of ABC/MBC (locoregionally recurrent not amenable to curative therapy or metastatic)
3. Patient with histologically and/or cytologically confirmed diagnosis of HR-positive (ER+ and/or PgR+), as well as HER2-negative breast cancer by local laboratory (HER2- by Immunohistochemistry [IHC], for borderline2+ Fluorescence In Situ Hybridization [FISH])
4. A separate signed patient ICF for Part A of the study must be obtained prior to any data collection and sample shipment to the central designated laboratory
5. Patient's tumor tissue (archival or fresh) is available to be sent to a central laboratory for PIK3CA testing. In case, tissue sample (archival or fresh) is not available or feasible, liquid biopsy may be allowed.

PART B:

1. Males (≥18 years of age), post-menopausal* females or pre-menopausal** females with ovarian ablation (as per physician decision).
2. Patients with confirmed diagnosis of ABC/MBC (locoregionally recurrent not amenable to curative therapy or metastatic) - for direct enrollment patients into Part B of the study.
3. Patient with histologically and/or cytologically confirmed diagnosis of HR-positive (ER+ and/or PgR+), as well as HER2-negative breast cancer by local laboratory (HER2- by Immunohistochemistry [IHC], for borderline2+ Fluorescence In Situ Hybridization [FISH]) - for direct enrollment patients into Part B of the study.
4. Participants with confirmed positive PIK3CA mutation status prior to study entry.
5. A separate signed ICF for Part B of the study must be obtained by all the patients, prior to any data collection, irrespective of patients who are being enrolled from Part A of the study or who are being enrolled directly into Part B of the study.
6. Physician decision to treat patients with alpelisib plus fulvestrant, according to the prescribing label and the local practicing guidelines.
7. Patient should be alpelisib treatment naïve.

Exclusion Criteria:

PART A:

1. Prior or current enrollment in any interventional clinical trial for ABC/MBC.

Part

PART B:

1. Patients' who had prior or current exposure to alpelisib or had prior or current exposure to any other PIK3CA inhibitor should be excluded.
2. Known hypersensitivity to alpelisib or fulvestrant, or to any of the excipients of alpelisib or fulvestrant.
3. Participant with type I or uncontrolled type II diabetes mellitus (HbA1c >7, [as per ADA/ACP guidelines 2020]).
4. Participant has a history of severe cutaneous reactions like Stevens-Johnson-Syndrome (SJS), Erythema Multiforme (EM), Toxic Epidermal Necrolysis (TEN), or Drug Reaction with Eosinophilia and Systemic Symptoms (DRESS).
5. Participant has documented pneumonitis/interstitial lung disease which is active and requiring treatment.
6. Participant with unresolved osteonecrosis of the jaw.
7. Participant reports history of acute pancreatitis within 1 year of screening or past medical history of chronic pancreatitis, major surgery, any relevant medical condition, gastrointestinal (GI) condition preventing absorption, Child Pugh score B or C etc.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PART A: males, post-menopausal women or pre-menopausal women who are receiving ovarian ablation PART B: patients who are PIK3CA mutation positive
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
PART A: Percentage of patients with tumors harboring a PIK3CA mutation | Baseline
  Defined as whether PIK3CA mutation is detected (positive or negative) after the enrollment of patient in Part A of the study.
  The mutation status should specify each 11 hotspots (C420R, E542K, E545A,E545D, E545G, E545K, Q546E, Q546R, H1047L, H1047R, and H1047Y)
PART B: Clinical Benefit Rate (CBR) as measured by RECIST 1.1 | Up to 24 months
  CBR defined as the proportion of patients with a best overall response of CR (complete response) or PR (partial disease), or an overall lesion response of stable disease (SD) or non-CR/non-PD (progressive disease) which lasts for a minimum time duration (with a default of at least 24 weeks in breast cancer studies). This should be evaluated as per RECIST v1.1. This endpoint measures signs of activity considering duration of disease stabilization

SECONDARY OUTCOMES:
PART A: Age at early stage (initial) disease, and advanced/metastatic disease diagnosis | Baseline
  Two sub-groups will be identified based on age as <75 years and ≥75 years for patient's data collection
PART A: Clinical characteristics of the disease at early (initial) stage of diagnosis- TNM staging | Baseline
  TNM staging will be collected
PART A: Clinical characteristics of the disease at early (initial) stage of diagnosis - receptor expression | Baseline
  Receptor expression can be:
  * ER: Estrogen Receptor
  * PgR: Progesterone Receptor
  * HER2: Human Epidermal Growth Factor Receptor 2
PART A: Clinical characteristics of advanced / metastatic disease stage - disease free interval (DFI) | Baseline
  Disease free interval (DFI) is defined as the interval from the completion of therapy to the diagnosis of recurrence
PART A: Clinical characteristics of advanced / metastatic disease stage - number of metastasis | Baseline
  At advanced / metastatic disease diagnosis number of metastasis will be collected
PART A: Clinical characteristics of advanced / metastatic disease stage - location of metastasis | Baseline
  At advanced / metastatic disease diagnosis location of metastasis will be collected
PART A: Clinical characteristics of advanced / metastatic disease stage - receptor expression | Baseline
  Receptor expression can be:
  * ER: Estrogen Receptor
  * PgR: Progesterone Receptor
  * HER2: Human Epidermal Growth Factor Receptor 2
PART A: Prior number of LoT for the advanced / metastatic disease | Baseline
  To identify the treatment patterns of prior therapies received for ABC/MBC, as available in the patient's medical record, prior number of Line of Therapy (LoT) for the advanced / metastatic disease will be collected
PART A: Prior treatment type | Baseline
  To identify the treatment patterns of prior therapies received for ABC/MBC, as available in the patient's medical record, prior treatment type (hormone alone, hormone with targeted therapy (TT), chemotherapy, etc.) will be collected
PART A: Prior treatment sequence by LoT | Baseline
  To identify the treatment patterns of prior therapies received for ABC/MBC, as available in the patient's medical record, prior treatment sequence by Line of Therapy (LoT) will be collected
PART A: Time to next treatment | Baseline
  To identify the treatment patterns of prior therapies received for ABC/MBC, as available in the patient's medical record, time to next treatment will be collected.
  Time to next treatment: defined as time gap between two Line of Therapy (LoT), as applicable
PART A: Reason (s) for discontinuation of prior therapy | Baseline
  To identify the treatment patterns of prior therapies received for ABC/MBC, as available in the patient's medical record, reason (s) for discontinuation of prior therapy will be collected
PART A: PIK3CA mutation positive patients not prescribed alpelisib | Baseline
  To identify the treatment patterns of prior therapies received for ABC/MBC, as available in the patient's medical record, PIK3CA mutation positive patients not prescribed alpelisib will be collected by reason
PART B: Progression Free Survival (PFS) by RECIST 1.1 | Up to 24 months
  Defined as the time from start of treatment with alpelisib plus fulvestrant (index date) to the date of the first documented progression or death due to any cause. If a patient has not had an event, PFS is censored at the date of last adequate tumor assessment.
PART B: Overall Response Rate (ORR) by RECIST 1.1 | Up to 24 months
  ORR is defined as the proportion of patients with best overall response of Complete Response (CR) or partial response (PR) evaluated based on local investigator's assessment according to RECIST 1.1
PARTB: Duration of response (DoR) by RECIST 1.1 | Up to 24 months
  Calculated as the time from the date of the first documented Complete Response (CR) or partial response (PR) per RECIST version 1.1.
PART B: Tolerability of alpelisib plus fulvestrant measured by adverse events (AEs) | Up to 24 months
PART B: Number of patients with laboratory abnormalities | Baseline, Up to 24 months
  The laboratory assessment will be recorded at baseline and during the study observation period based on changes in Grade of laboratory abnormality.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- India (21):
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Guwahati, Assam
  - Novartis Investigative Site, Kochi, Kerala
  - Novartis Investigative Site, Bhopal, Madhya Pradesh
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Bhubaneshwar, Odisha
  - Novartis Investigative Site, Bhubaneswar, Odisha
  - Novartis Investigative Site, Chandigarh, Punjab
  - Novartis Investigative Site, Ludhiana, Punjab
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, Sherilingampally, Telangana
  - Novartis Investigative Site, Howrah, West Bengal
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, Ahmedabad
  - Novartis Investigative Site, Kanpur
  - Novartis Investigative Site, Kolkata
  - Novartis Investigative Site, Puducherry
  - Novartis Investigative Site, Udaipur

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to study results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18414